CLINICAL TRIAL: NCT01549678
Title: Effect of Plantar Fasciitis Foot Insole
Brief Title: Plantar Fasciitis Foot Insole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Hilda Alcantara Veiga de Oliveira, Effect of Fasciitis Plantar Foot Insoles, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1349/09
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2010-11

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis; foot pain; insoles; foot function; electronic baropodometer; plantar pressure; gait analysis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention foot orthoses (Experimental): Ethyl Vinil Acetate EVA insole shaped in the cast of the patient's foot.
  Interventions: Other: Total contact insole
- Placebo insole (Placebo Comparator): EVA flat insole.
  Interventions: Other: placebo insole

INTERVENTIONS:
Other: Total contact insole — EVA insole shaped on patient´s foot.
  Other Names: Intervention group
  Arms: Intervention foot orthoses
Other: placebo insole — EVA insole flat
  Other Names: Placebo group
  Arms: Placebo insole

SUMMARY:
The hypothesis to be tested is that the use of total contact insoles for six months reduces foot pain, improves function and quality of life of patients diagnosed with plantar fasciitis.

DETAILED DESCRIPTION:
Patients diagnosed with plantar fasciitis, foot pain with VAS between 3 - 8 for walk, over 18 years, regardless of gender who agreed to participate and signing the consent form. Pacietes We excluded patients with other symptomatic lower limb musculoskeletal diseases, diabetes mellitus, rigid deformities in the feet, which made use of insoles, physiotherapy or injections in feet and ankles in the last three months, and previous surgery or planned within the next twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a diagnosis of PF and foot pain while walking ranging from 3 to 8 points on a 10-point pain scale were analyzed

Exclusion Criteria:

* Patients with other musculoskeletal conditions in symptomatic lower limbs, inflammatory conditions of the central or peripheral nervous systems, diabetes mellitus or an inability to walk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-04 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale of pain in feet during walking (VAS) | Six months
  Assessing pain in the feet during walking through a visual analog scale from 0 to 10

SECONDARY OUTCOMES:
FFI | 6 months
  Questionaire of function of the foot
FHSQ-Br | 6 months
  Foot Health Status Questionaire
Visual analog scale of pain in feet at reset (VAS) | 6 months
  Assessing pain in the feet at reset through a visual analog scale from 0 to 10
6-MINUTE WALK TEST | 6 months
  Assess functional capacity
SF-36 | 12 months
  Assess functional capacity
Likert scale | 6 months
  Likert scale by patients
Baropodometric tests | 6 months
  Evaluates charge gistribution in the feet and gait variables
Time use of insole | 6 months
  Control use of insole

CONTACTS AND LOCATIONS:
Overall Officials: Hilda PT Oliveira, Principal Investigator — Federal University of São Paulo; Anamaria PT Jones, PHD, Study Director — Federal University of São Paulo; Jamil MD Natour, PHD, Study Chair — Chief of Rheumatology, Federal
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil